CLINICAL TRIAL: NCT02433184
Title: A Prospective, Single-centre, Randomised Study Evaluating the Clinical, Imaging and Immunological Depth of Remission Achieved by Very Early Versus Delayed Etanercept in Patients With Rheumatoid Arthritis
Brief Title: Very Early Versus Delayed Etanercept in Patients With RA
Acronym: VEDERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Maya Buch, NIHR Clinician Scientist, Senior Lecturer/Honorary Consultant Rheumatologist, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR10/9592
Record Dates: First submitted 2015-04-23; First posted 2015-05-04 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Etanercept; treat to target; Disease Modifying Antirheumatic Drugs (DMARDs)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate; Sulfasalazine; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etanercept (Experimental): Treatment Arm 1 will receive etanercept and methotrexate combination therapy administered for a total duration of 48 weeks.
  Interventions: Drug: Etanercept; Drug: Methotrexate
- Methotrexate-treat to target (Active Comparator): Treatment Arm 2 will receive initial methotrexate monotherapy with adoption of a treat to target protocol (standard care involving monthly DAS28-ESR assessment with escalation to combination sDMARD therapy if not achieving LDA at, or after, 8 weeks) and step-up to etanercept and methotrexate at 24 weeks if failing to achieve clinical remission
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Hydroxychloroquine; Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept will be administered subcutaneously at a dose of 50 mg weekly and will be discontinued at the primary endpoint (48 weeks).
  Arms: Etanercept
Drug: Methotrexate — Methotrexate will be administered orally at a starting dose of 15 mg and will be increased to 25mg weekly at 2 weeks.
  Arms: Methotrexate-treat to target
Drug: Sulfasalazine — Sulfasalazine will be added at weeks 8,12,16 or 20 if the subject fails to achieve low disease activity, administered orally at a dose of 1g twice daily. Will be discontinued if starting etanercept at 24 weeks.
  Arms: Methotrexate-treat to target
Drug: Hydroxychloroquine — Hydroxychloroquine will be added at weeks 8,12,16 or 20 if the subject fails to achieve low disease activity, administered at a dose of 200mg daily. Will be discontinued if starting etanercept at 24 weeks.
  Arms: Methotrexate-treat to target
Drug: Etanercept — Etanercept will be added at 24 weeks, if a subject fails to achieve clinical remission,at a dose of 50 mg weekly and will be discontinued at 48 weeks with the exception of those patients who are eligible to continue according to local prescribing guidelines (NICE guidelines)
  Arms: Methotrexate-treat to target
Drug: Methotrexate — Methotrexate will be administered orally at a starting dose of 15 mg weekly, increasing to 20mg and 25mg weekly at weeks 4 and 8 respectively.
  Arms: Etanercept

SUMMARY:
The main aim of the study is to determine whether TNFi instituted as first-line therapy in early RA confers better outcomes (clinical, structural and immunological) compared to delayed TNFi start; implying particular dominance of TNF in early disease, a changing role of TNF with disease duration and hence, confirmation of a biological window of opportunity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 18 and 80 years.
* Diagnosis of rheumatoid arthritis (new 2010 ACR/EULAR RA classification criteria).
* Symptom onset within the preceding 12 months.
* Patients with active RA at baseline: clinical evidence of synovitis (or imaging evidence of synovitis in cases of uncertainty/subclinical disease) in hand and/or wrist joints evaluable by ultrasound and MRI, and DAS28-ESR>3.2.
* Seropositivity for anti-citrullinated peptide antibody (ACPA) and/or rheumatoid factor. If ACPA and rheumatoid factor are both negative, presence of power Doppler in at least 1 joint on ultrasound imaging.
* DMARD-naive (with the exception of previous exposure to hydroxychloroquine for an indication other than RA).
* All male and female subjects biologically capable of having children must agree to use a reliable method of contraception for the duration of the study and 24 weeks after the end of the study period. Acceptable methods of contraception are surgical sterilisation, oral, implantable or injectable hormonal methods, intrauterine devices or barrier contraceptives.

Exclusion Criteria:

* Previous treatment with DMARDs for the management of RA.
* Intramuscular or intra-articular (of non-target joint) corticosteroid within 28 days of the screening visit; intra-articular steroid of the chosen target joint within 12 weeks of screening.
* Oral steroid of greater than 10mg prednisolone daily, or change in oral steroid dose within 28 days of study drug initiation at the baseline visit.
* Use (including use as required) of more than one NSAID, change in NSAID or change in dose of NSAID within 28 days of the baseline visit.
* Contraindications to MRI (e.g. pacemaker) or unable or unwilling to attend for all imaging assessments. In patients with previous penetrating trauma to the eye, or patients at high risk of previous metal foreign body injury to the eye (e.g. welding), skull x-ray will be performed; these patients may be included in the absence of residual metal fragments on x-ray.
* Pregnancy or breastfeeding.
* Other contraindications to TNFi as determined by local prescribing guidelines and physician discretion, including:

  * Active infection, open leg ulcers, previously infected prosthetic joint (unless completely removed), septic arthritis in last year, HIV, Hepatitis B or Hepatitis C carriers, previous malignancy within 10 years (except basal cell carcinoma), severe heart failure (New York Heart Association grade 3 or more), any history of demyelinating disease, uncontrolled diabetes, pulmonary fibrosis, bronchiectasis, previous PUVA therapy (of >1000 Joules), history of TB or evidence of latent TB on chest x-ray/TB testing (in the latter event, a patient may be included if treated with isoniazid and pyridoxine one month before starting the study and for a further 6 months whilst on study treatments).
* History of other significant medical conditions, including:

  * Severe pulmonary disease, defined as requiring previous hospital admission or supplemental oxygen.
  * Active or severe cardiovascular disease: uncontrolled hypertension, myocardial infarction within 12 months of screening, unstable angina within 6 months of screening.
  * Other immunodeficiency disorders.
  * Connective tissue diseases, e.g. primary Sjogren's syndrome, systemic sclerosis, systemic lupus erythematosus, polymyositis.
  * Psoriasis.
  * Renal impairment (creatinine ≥ 175µmol/L).
  * Blood disorders: neutropenia (neutrophils < 2.0 x 109/L), thrombocytopenia (platelets < 125 x 109/L), or anaemia (haemoglobin < 8 g/dL).
  * Abnormal liver function (alanine transaminase, ALT > 3 x upper limit of normal).
* Planned surgery within the study period which is expected to require omission of any study medication of 28 days or more.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Clinical remission | 48 weeks
  Proportion of patients that achieve clinical remission (Disease activity Score, DAS28 <2.6) at 48 weeks, following either treatment strategy.

SECONDARY OUTCOMES:
Change in MRI synovitis | baseline and week 48
  Change in MRI synovitis between baseline and 48 weeks.
CDAI (clinical disease activity index) | weeks 12, 24, 48 and 96
  Change in CDAI score from baseline at weeks 12, 24, 48 and 96
SDAI (simplified disease activity index) | weeks 12, 24, 48 and 96
  Change in SDAI score from baseline at weeks 12, 24, 36 & 48.
ACR(American College of Rheumatology) response scores | weeks 12, 24, 48 and 96
  ACR response score from baseline at weeks 12, 24, 48 and 96
EULAR(European League Against Rheumatism)response criteria | weeks 12, 24, 48 and 96
  EULAR response score from baseline
Physical function, assessed by HAQ(health assessment questionnaire) | weeks 12, 24, 48 and 96
Quality of life scores assessed by RA-QoL(RA quality of life questionnaire) | weeks 12, 24, 48 and 96
Work instability, assessed by RA-WIS(RA work instability questionnaire) | weeks 12, 24, 48 and 96
HRUS (High Resolution Ultrasound) | weeks 0, 12, 24 and 48
  Change in HRUS from baseline
Radiographic scores | weeks 48 and 96
  Change in joint damage assessed by modified Sharp score.
Immunological parameters in blood sample | weeks 0, 12, 24 and 48
  Change in immunological markers of inflammation between baseline and weeks 12, 24 and 48.
Immunological parameters in synovial tissue | weeks 0, 24, +/- 48
  Change in immunological markers of inflammation between baseline and weeks 24 and 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Rheumatic & Musculoskeletal Medicine, Chapel Allerton Hospital, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Emery P, Horton S, Dumitru RB, Naraghi K, van der Heijde D, Wakefield RJ, Hensor EMA, Buch MH. Pragmatic randomised controlled trial of very early etanercept and MTX versus MTX with delayed etanercept in RA: the VEDERA trial. Ann Rheum Dis. 2020 Apr;79(4):464-471. doi: 10.1136/annrheumdis-2019-216539. Epub 2020 Jan 29. PMID 31996367
- [Derived] Dumitru RB, Horton S, Hodgson R, Wakefield RJ, Hensor EMA, Emery P, Buch MH. A prospective, single-centre, randomised study evaluating the clinical, imaging and immunological depth of remission achieved by very early versus delayed Etanercept in patients with Rheumatoid Arthritis (VEDERA). BMC Musculoskelet Disord. 2016 Feb 5;17:61. doi: 10.1186/s12891-016-0915-0. PMID 26847108